CLINICAL TRIAL: NCT07111247
Title: Insights in Endocervical Mucus Secretion
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Leo Han, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00028821; R01HD115770-01A1 (NIH)
Record Dates: First submitted 2025-07-28; First posted 2025-08-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cervical Mucus
MeSH Terms: interventions — relugolix

STUDY DESIGN:
Intervention Model Description: All participants will receive Relugolix for 10 days starting at the midluteal time point
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Relugolix (Experimental): Participants will take Reugolix for 10 days starting at the midluteal time point (6-9 days after "high fertility" based on ovulation test)
  Interventions: Drug: Gonadotropin Releasing Hormone Antagonists Relugolix

INTERVENTIONS:
Drug: Gonadotropin Releasing Hormone Antagonists Relugolix — Gonadotropin releasing hormone antagonist (gnRH) taken for 10 days starting during the midluteal phase.

SUMMARY:
Single arm interventional study looking at biological outcomes at 4 time points throughout the cycle before and after taking an oral gonadotropin-releasing hormone antagonist (gnRH). Samples of whole blood, endocervical mucus, endocervical biopsy, and vaginal swab will be collected.

DETAILED DESCRIPTION:
This study will enroll participants and obtain biological samples at 4 time points. The study will begin on the first day of menstruation following enrollment. Patients will monitor for peri-ovulation using an ovulation test that monitors for urinary metabolites for luteinizing hormone (LH). At the midluteal time point for sampling (days 6-9 after "high fertility" on ovulation test) subjects will begin taking an oral gonadotropin-releasing hormone antagonist (gnRH) (relugolix) for 10 days. Samples of whole blood, endocervical mucus, endocervical biopsy, and vaginal swab will be collected during the early follicular phase (3-5 days following the start of menstruation), peri-ovulation (9-14 days following the start of menstruation based on estriol glucuronide (E3G) urinary metabolite), mid-luteal (6-9 days following mid-cycle draw), and upon stoppage of relugolix (9-11 days following relugolix initiation).

ELIGIBILITY:
Inclusion Criteria:

* Normal menstrual cycles of 25-35 days in length for at least the previous 3 cycles
* BMI >18 and <35
* Serum p4 >= 3 ng/ml on single sample collected between days 18-25 of self-reported menstrual cycle
* Flexible schedule allowing blood draws on less than 48 hour notice
* In good general health
* Commit to using non-hormonal contraceptive methods without spermicide during study period except those prescribed in the experimental protocol
* No objections to taking study drugs
* No objections to refraining from intercourse the night before any sampling and willing to use condoms during vaginal intercourse

Exclusion Criteria:

* Oral contraceptive use or other hormone supplement within the preceding 2 months
* Current cervical infection
* Evidence of abnormal cervical cytology
* Use of any IUD for contraception
* Long-acting hormonal contraceptive use in the past 12 months (e.g., Depo-Provera)
* Contraindications to study drugs
* Current or past pregnancy within the previous 6 months or currently trying to conceive
* Desiring to conceive in the next 8 months
* Breastfeeding in the past 2 months
* Diagnosed diabetes or metabolic syndrome
* Diagnosed Polycystic Ovary Syndrome
* History of, or self-reported, substance abuse
* Smoker
* Previous infertility treatment excluding male factor issues
* Use of an investigational drug within the past 2 months
* History of excisional or ablative treatment procedure on cervix (i.e., LEEP, Cryotherapy, Cold Knife Cone)
* Current treatment for a vaginal infection such as bacterial vaginosis
* History of venous thromboembolism (VTE) or inherited thrombophilias

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Cervical mucus scores | Cervical mucus will be collected and compared across 4 time points during the menstrual cycle (follicular [3-5 days following start of menses], ovulatory, luteal, ovarian suppression [9-11 days following Relugolix initiation])
  Average cervical mucus scores at each study time point
Single cell transcriptome analysis | Measured and compared across 4 time points during the menstrual cycle (follicular [3-5 days following start of menses], ovulatory, luteal, ovarian suppression [9-11 days following Relugolix initiation])
  Single cell transcriptome analysis comparing changes across menstrual time points
Proteomic analysis | Measured and compared across 4 time points during the menstrual cycle (follicular [3-5 days following start of menses], ovulatory, luteal, ovarian suppression [9-11 days following Relugolix initiation])
  Proteomic analysis of mucus including Mucin concentration

CONTACTS AND LOCATIONS:
Overall Officials: Leo Han, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States